CLINICAL TRIAL: NCT01851993
Title: Effects of Inhaled Ondansetron on Perceived Respiratory Discomfort (Dyspnea) During Exercise in the Presence of External Thoracic Restriction
Brief Title: Inhaled Ondansetron & Dyspnea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A02-M16-13B Ondansetron
Record Dates: First submitted 2013-05-07; First posted 2013-05-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Dyspnea
Keywords: Ondansetron; Exercise
MeSH Terms: conditions — Dyspnea; Motor Activity | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled Ondansetron (8 mg) (Experimental): Single-dose inhalation of nebulized ondansetron (8 mg)
  Interventions: Drug: Ondansetron
- Inhaled 0.9% saline placebo (Placebo Comparator): Single-dose inhalation of 0.9% saline placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron
  Arms: Inhaled Ondansetron (8 mg)
Drug: Placebo — 0.9% saline
  Arms: Inhaled 0.9% saline placebo

SUMMARY:
"Dyspnea" refers to the awareness of breathing discomfort that is typically experienced during exercise in health and disease. In various participant populations, dyspnea is a predictor of disability and death; and contributes to exercise intolerance and an adverse health-related quality-of-life. It follows that alleviating dyspnea and improving exercise tolerance are among the principal goals of disease management. Nevertheless, the effective management of dyspnea and activity-limitation remains an elusive goal for many healthcare providers and current strategies aimed at reversing the underlying chronic disease are only partially successful in this regard. Thus, research aimed at identifying dyspnea-specific medications to complement existing therapies for the management of exertional symptoms is timely and clinically relevant. The purpose of this study is to test the hypothesis that single-dose inhalation of nebulized ondansetron (a serotonin 5-HT3 receptor antagonist) will improve the perception of dyspnea during strenuous exercise in health, young men. To this end, the investigators will compare the effects of inhaled 0.9% saline placebo and inhaled ondansetron (8 mg) on detailed assessments of neural respiratory drive (diaphragm EMG), ventilation, breathing pattern, dynamic operating lung volumes, contractile respiratory muscle function, cardio-metabolic function and dyspnea (sensory intensity and affective responses) during symptom-limited, high-intensity, constant-work-rate cycle exercise testing in healthy, men aged 20-40 years.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 20-40 years
* FEV1 ≥80% predicted
* FEV1/FVC >70%

Exclusion Criteria:

* Current or ex-smoker
* Body Mass Index <18.5 or >30 kg/m2
* History of cardiovascular, vascular, respiratory, renal, liver, musculoskeletal, endocrine, neuromuscular and/or metabolic disease/dysfunction.
* Taking doctor prescribed medications
* Allergy to latex
* Allergy to lidocaine or its "caine" derivatives

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sensory Intensity (Borg 0-10 scale) ratings of dyspnea at isotime | Participants will be followed until all study visits are complete, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University, Montreal, Quebec, Canada

REFERENCES:
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl